CLINICAL TRIAL: NCT04147936
Title: A 12-Week, Single-Blind, Placebo-Controlled, Randomized Study to Evaluate the Safety, Tolerability, and Physiological Regulation of an Amino Acid Food Product, AXA1665, in Subjects With Mild and Moderate Hepatic Insufficiency
Brief Title: Study of the Safety and Tolerability of AXA1665 in Subjects With Mild and Moderate Hepatic Insufficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Axcella Health, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: AXA1665-002
Record Dates: First submitted 2019-10-21; First posted 2019-11-01 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Hepatic Insufficiency
Keywords: Amino acids, food study
MeSH Terms: conditions — Hepatic Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AXA1665 29.4g (Active Comparator): Dietary Supplement: AXA1665 Amino acids, food study
  Interventions: Dietary Supplement: AXA1665
- AXA1665 53.9 g (Active Comparator): Dietary Supplement: AXA1665 Amino acids, food study
  Interventions: Dietary Supplement: AXA1665
- Placebo 29.4 g (Placebo Comparator): Dietary Supplement: Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: AXA1665 — Dietary supplement: AXA1665
  Arms: AXA1665 29.4g; AXA1665 53.9 g
Dietary Supplement: Placebo — Placebo
  Arms: Placebo 29.4 g

SUMMARY:
This is a randomized, single blind study to determine whether AXA1665, a composition of naturally occuring amino acids, is well tolerated in subjects with mild and moderate hepatic insufficiency. Study will also examine how the food product may influence the biology in muscle which will be assessed using magnetic resonance imaging (MRI) and other functional assessments such as strength, balance and cognition as part of a comprehensive physical/neurological exam. Changes in blood biomarkers of inflammation will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in the study and provide written informed consent
* Male and female adults aged > 18 years
* Child-Pugh score ≤9 (i.e. Child-Pugh class A or B)
* Liver Frailty Index (LFI) of ≥3.6
* Willing and able to engage in 30 minutes of walking/physical activity at least 3 days per week

Exclusion Criteria:

* Hospitalization for any complication of cirrhosis or taking new medications intended to treat hepatic encephalopathy within 2 months prior to Screening or any hospitalization for any cause/reason within 30 days prior to Screening
* Prior history or presence of a transjugular intrahepatic portal systemic shunt (TIPS)
* Current or history of significant alcohol consumption
* Other poorly controlled medical condition [e.g., renal disease with an estimated glomerular filtration rate (GFR) <60 mL/min/1.73m2)
* Known sensitivity and/or history of clinically significant food intolerance/allergies to proteins (including whey, soy, casein, amino acids, etc.)
* Any extreme or unbalanced diet such as Ketogenic, Atkins, Paleo, Vegan, etc.
* Unable or unwilling to adhere to contraception requirements
* Any contraindications to a MRI scan
* Any other condition that, in the opinion of the Investigator, renders the subject at risk for compliance, compromises the well-being of the subject, or hinders study completion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-30 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-06-24 (Actual)

PRIMARY OUTCOMES:
Incidence of study product emergent adverse events (AEs) and serious adverse events (SAEs) | Baseline to Week 12

SECONDARY OUTCOMES:
Change in muscle mass by MRI | Baseline to Week 12
Change in Fischer's ratio [measured by ratio of branched-chain amino acids (leucine, valine, isoleucine) to aromatic amino acids (phenylalanine, tyrosine)] | Baseline to Week 12
Change in plasma ammonia | Baseline to Week 12
Change in blood urea nitrogen concentration | Baseline to Week 12
Change in creatinine concentration | Baseline to Week 12
Change in gait speed | Baseline to Week 12
Change in Liver Frailty Index | Baseline to Week 12
Change in overall physical activity (measured by actigraphy watch) | Baseline to Week 12
Change in cognitive function measured by the Psychometric Hepatic Encephalopathy Score (PHES) | Baseline to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Arun J Sanyal, MD, Principal Investigator — Virginia Commonwealth University
Locations (11):
- United States (11):
  - Catalina Research Institute, LLC, Montclair, California
  - Orange County Research Center, Tustin, California
  - Panax Clinical Research, Miami Lakes, Florida
  - OMEGA Research Maitland, LCC, Orlando, Florida
  - Avita Clinical Research, Tampa, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Indiana University Health, Indianapolis, Indiana
  - Delta Research Partners, Bastrop, Louisiana
  - UPMC Center for Liver Disease, Pittsburgh, Pennsylvania
  - Texas Liver Institute, San Antonio, Texas
  - Virginia Commonwealth University, Richmond, Virginia